CLINICAL TRIAL: NCT05792553
Title: Effects of Tongue Tamers and Customized Bonded Spurs as an Early Treatment of Anterior Open Bite: A Randomized Clinical Study
Brief Title: Effects of Tongue Tamers as an Early Treatment of Anterior Open Bite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Safa Basiouny Alawy, Lecturer of Orthodontics, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #R-ORTH-2-23-5
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Tongue Habits; Open Bite
Keywords: open bite; tongue thrust; habit breaking appliance
MeSH Terms: conditions — Tongue Habits; Open Bite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group I: bonded tongue tamers (Experimental): 25 cases with anterior open bite will be treated using bonded tongue tamers
  Interventions: Device: bonded tongue tamers
- group II: customized bonded spurs (Experimental): 25 cases with anterior open bite will be treated using customized bonded spurs
  Interventions: Device: customized bonded spurs
- group III: conventional fixed palatal spurs (Active Comparator): 25 cases with anterior open bite will be treated using conventional fixed palatal spurs
  Interventions: Device: conventional fixed palatal spurs

INTERVENTIONS:
Device: bonded tongue tamers — Enamel surface will be treated initially with 37% phosphoric acid for 30 seconds then tongue tamers will be bonded to the palatal/lingual surface of upper and lower central incisors
  Arms: group I: bonded tongue tamers
Device: customized bonded spurs — Composite restoration will be used to fabricate the customized bonded spurs with sharp ends and 3 mm in length.
  Arms: group II: customized bonded spurs
Device: conventional fixed palatal spurs — conventional fixed palatal spurs will be fabricated by taking impression after band selection, then the spurs appliance will be fabricated from 0.9 mm stainless steel wire and soldered to the bands bilaterally.
  Arms: group III: conventional fixed palatal spurs

SUMMARY:
Anterior open bite (AOB) is a malocclusion that causes aesthetic, speech, feeding, and psychological concerns, emphasizing the significance of beginning treatment as soon as possible to correct the disorder. The main etiological determinants of AOB include finger-sucking, pacifiers, and oral habits; hence, it is vital to use interceptive treatments focused on correcting and increasing bite stability during childhood to avoid the need for advanced therapy

ELIGIBILITY:
Inclusion Criteria:

* male or female patients in early mixed dentition period with age range 7-9 years
* dental anterior open bite equal to or greater than 1 mm,
* class I malocclusion
* clinical signs of anterior tongue thrusting.

Exclusion Criteria:

* Patients with skeletal open bite
* posterior crossbite
* tooth agenesis or loss of permanent teeth
* crowding,
* systemic diseases

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Change of the anterior open bite | 3 months
  Measuring method: Digital caliper Measuring unit: Binary (+/-)

SECONDARY OUTCOMES:
cephalometric variables | 3 months
  cephalometric variables including SNA°, SNB°, ANB°, FMA°, U1/FHP°, L1/GoGn°, and overjet will be analyzed pre- and post- treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

REFERENCES:
- [Derived] Alawy SB, El-Desouky SS, Kabbash IA, Hadwa SM. Effects of tongue tamers and customized bonded spurs as an early treatment of anterior open bite: a randomized clinical study. BMC Oral Health. 2025 Jan 16;25(1):76. doi: 10.1186/s12903-024-05389-x. PMID 39819458